CLINICAL TRIAL: NCT05400590
Title: Comparison of the Healing Properties on Corneal Cells of Groth Factor-enriched Plasma and Autologous Serum From Aniridia Patients
Acronym: CICASAND
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: DGT_2022_2; 2022-A00259-34 (Other: IDRCB)
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Aniridia
Keywords: Growth factor rich plasma; Conjunctival impression
MeSH Terms: conditions — Aniridia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case patients with aniridia
  Interventions: Procedure: Peripheral venous blood sample; Procedure: Conjunctival impression
- Control patients without aniridia
  Interventions: Procedure: Peripheral venous blood sample; Procedure: Conjunctival impression

INTERVENTIONS:
Procedure: Peripheral venous blood sample — 2.5% of body weight
Procedure: Conjunctival impression — Collection of the most superficial conjunctival epithelial cells (desquamating) in a non- or minimally invasive, quick and almost painless way, for a biological analysis of ocular surface diseases. Application of a filter paper on the bulbar conjunctiva, under local anesthesia.

SUMMARY:
Keratopathy of patients with aniridia leads to epithelial scarring disorders and a progressive clouding of the cornea linked to this abnormal healing (fibrosis). Treatment with autologous serum is usually undertaken to promote epithelial healing.

However, autologous serum does not prevent the formation of fibrosis, whereas growth factor-rich plasma appears to be associated with a reduction in the in vitro expression of fibrosis markers. This study seeks to compare the in vitro healing and anti-fibrotic properties of autologous serum and growth factor rich plasma from aniridia patients and healthy controls.

DETAILED DESCRIPTION:
Blood collection from aniridia patients and healthy controls, half of which will be used to make autologous serum and the other half to make growth factor rich plasma, used for in vitro studies.

A conjunctival impression will also be taken at the inclusion of the patients.

ELIGIBILITY:
Inclusion Criteria:

For patients with aniridia:

* With aniridia
* Patient weighing more than 43 kg
* If the patient is being treated with autologous serum, a delay of 8 weeks after the last blood collection
* If a blood donation has been made, a delay of 8 weeks must be respected after the last donation

For controls:

* Non-aniridia (no clinical signs)
* Weighing more than 43 kg
* Matched to a case for sex and age +/-10 years
* No known diabetes
* If a blood donation has been made, a delay of 8 weeks must be respected after the latter

Exclusion Criteria:

* Insufficient sample volume
* No conjunctival print
* HBV, HCV, HIV serology positive
* Aniridia not genetically confirmed for cases For each patient excluded, a new patient will be included in order to maintain the number of patients required for data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aniridia patients and controls without aniridia
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
In vitro comparison of the corneal cell healing properties of autologous serum and plasma enriched with growth factors from blood of aniridia patients | Sampling done at baseline
  The corneal cell healing properties are evaluated by the time to reach confluence (number of hours) of epithelial cells, using a standardized wound healing assay (Incucyte, Essenbioscience). The corneal cell healing properties will be comparated between autologous serum, and plasma enriched with growth factors from blood of aniridia patients

CONTACTS AND LOCATIONS:
Overall Officials: Eric GABISON, Study Chair — Hôpital Fondation A. de Rothschild; Damien GUINDOLET, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France